CLINICAL TRIAL: NCT03609112
Title: Neurocognitive Risks in Children With Solid Tumors
Acronym: RISK-N
Status: Recruiting | Type: Observational
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A00924-43; 2014/2127 (Other: CSET number)
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor in Children
MeSH Terms: interventions — The Brief Resilience Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients treated for a brain tumor: As part of their usual follow-up, these patients have neuropsychological evaluations following their treatment. A complete neuropsychological evaluation will therefore be performed as part of their usual follow-up during the inclusion period of this study and only the data from this evaluation will be taken into account for the statistical analysis of this study.
  Interventions: Other: The WISC-V; Other: The NEPSY-II; Other: The Child Executive Function Evaluation Battery CEF; Other: The "CONNERS 3 long version"; Other: The "BRIEF"; Other: The "PEDS-QL quality of life"; Other: The 'fatigue' version of the PEDS-QL (Tessier et al., 2009: parent and child-adolescent version for the brain tumour cohort); Other: The Family Functioning Inventory FAD)
- Patients treated for a non-cerebral tumor: A single neuropsychological assessment will be proposed to these patients after the end of treatment and during the inclusion period of this study. This evaluation will be carried out during a visit to Gustave Roussy as part of their usual follow-up. If on the occasion of this evaluation, cognitive disorders or psychological disorders were highlighted, a neuropsychological and / or psychological follow-up would be proposed.
  Interventions: Other: The WISC-V; Other: The Child Executive Function Evaluation Battery CEF; Other: The "CONNERS 3 long version"; Other: The "BRIEF"; Other: The Family Functioning Inventory FAD); Other: The 'fatigue' version of the PEDS-QL (Tessier et al., 2009: child version for the extra-cerebral tumour cohort)
- Patients who received Methotrexate: Methotrexate is used in the treatment of certain brain tumors as in that of non-cerebral tumors. Some of these patients, particularly those who have had neurological complications with methotrexate, will already have longitudinal neuropsychological follow-up as part of their usual follow-up. For these patients, only one complete neuropsychological assessment will be performed during the inclusion period and will be considered for statistical analysis.
  For patients in the course of treatment with methotrexate, during the period of inclusion of this study, a longitudinal follow-up will be carried out with neuropsychological evaluations close and successive at the time of their coming to Gustave Roussy within the usual framework of their care.
  Interventions: Other: The WISC-V; Other: The Child Executive Function Evaluation Battery CEF; Other: The "CONNERS 3 long version"; Other: The "BRIEF"; Other: The Family Functioning Inventory FAD); Other: The 'fatigue' version of the PEDS-QL (Tessier et al., 2009: child version for the extra-cerebral tumour cohort)

INTERVENTIONS:
Other: The WISC-V — The WISC-V (Weschler, 2016) which is measured with several indices: Verbal Comprehension Index (VCI), Visual Spatial Index (VSI), Working Memory Index (WMI), Fluid Reasoning Index (FRI), Processing Speed Index (PSI), and Full Scale IS (FSIQ).
Other: The NEPSY-II — The NEPSY-II (Korkman et al., 2012). The Narrative Memory subtest is designed to assess verbal memory using organised language material.
  Groups: Patients treated for a brain tumor
Other: The Child Executive Function Evaluation Battery CEF — The Child Executive Function Evaluation Battery CEF (Roy et al., 2021), which aims to evaluate the four main components of executive function (inhibition, working memory, flexibility and planning).
Other: The "CONNERS 3 long version" — The " CONNERS 3 long version " (Conners, 2008), which assesses attentional skills by means of a questionnaire to be completed by parents.
Other: The "BRIEF" — The 'BRIEF' (Gioia et al., 2013; parent version, teacher version), which is a behavioural evaluation inventory of executive functions completed by parents and teachers and which makes it possible to determine whether the child has, for example, difficulties with organisation, planning or behavioural regulation.
Other: The "PEDS-QL quality of life" — The "PEDS-QL quality of life" (Tessier et al., 2009) that will be completed by the parents and the patient concerns the day to- day functioning of the child (in school, relationships to others, physical abilities and emotional state).
  Groups: Patients treated for a brain tumor
Other: The 'fatigue' version of the PEDS-QL (Tessier et al., 2009: parent and child-adolescent version for the brain tumour cohort) — The 'fatigue' version of the PEDS-QL (Tessier et al., 2009: parent and child-adolescent version for the brain tumour cohort) which assesses fatigue in everyday life.
  Groups: Patients treated for a brain tumor
Other: The Family Functioning Inventory FAD) — The Family Functioning Inventory FAD (Speranza et al., 2006) is used to assess the family functioning of the child and his/her family. The short version is used as an indicator of general functioning.
Other: The 'fatigue' version of the PEDS-QL (Tessier et al., 2009: child version for the extra-cerebral tumour cohort) — The 'fatigue' version of the PEDS-QL (Tessier et al., 2009: child version for the extra-cerebral tumour cohort) which assesses fatigue in everyday life.
  Groups: Patients treated for a non-cerebral tumor; Patients who received Methotrexate

SUMMARY:
The survival rate of children with cancer has improved significantly in recent years thanks to the progress of different therapies. The neurocognitive sequelae related to treatments and illness are more or less well known. Four factors seem to be associated with neurocognitive sequelae: treatment, the tumor itself, environmental factors like the socio-economic status of parents and biological factors.

Main purpose of the study is to establish a score to assess the risk of neurocognitive sequelae in these children based on these factors (treatment, tumor, and environmental factors)

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 6 to 16 years and 11 months during the study period
* Type of pathology: solid tumor
* Place of treatment and follow-up: Gustave Roussy
* Minimum time from the end of the initial treatment:
* For patients who have not received treatment with methotrexate: 6 months
* For patients being treated with methotrexate: none
* Obtaining the non-opposition of parents / legal representatives
* Affiliation to a social security scheme.

Exclusion Criteria:

* Patients with other pathologies associated with mental retardation (autism, genetic syndrome ...)
* Patients lost to follow-up
* Deceased patients
* Patients treated for a pathology whose prognosis is involved in the very short term (infiltrating glioma of the brainstem, recurrence of the pathology during treatment)
* Non-French speaking patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient aged 6 to 16 years and 11 months during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of possible neurocognitive deficits according to the pathology and treatments received. | Up to 60 months
Univariate analysis to identify risk factors related to cognitive disorders. | Up to 60 months
Multiple regression analysis to determine the most significant risk factors and examine the interactions between these factors. | Up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided